CLINICAL TRIAL: NCT06717048
Title: An Exploratory Study on the Minimum Power and Frequency of Repeated Low-level Red-light to Effectively Control Myopia Progression
Brief Title: Minimum Power and Frequency of Repeated Low-level Red-light to Effectively Control Myopia Progression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RLPT-SEPTC-2024
Record Dates: First submitted 2024-11-03; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Myopia; Refractive Error - Myopia; Choroidal Thickness; Retina
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Red light: 2.0 mW/twice daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 2.0 mW/once daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 1.0 mW/twice daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 1.0 mW/once daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 0.5 mW/twice daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 0.5 mW/once daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 0.3 mW/twice daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red light: 0.3 mW/once daily (Experimental)
  Interventions: Device: Repeated Low-level Red-light
- Red LED: twice daily (Sham Comparator)
  Interventions: Device: Red LED

INTERVENTIONS:
Device: Repeated Low-level Red-light — In addition to single vision spectacle lenses (SVS) with power for correcting distance refraction, the subjects used the prescribed power low-intensity red light treatment instrument for the prescribed number of treatments from Monday to Friday, with a 3-minute interval of 4 hours.
  Arms: Red light: 0.3 mW/once daily; Red light: 0.3 mW/twice daily; Red light: 0.5 mW/once daily; Red light: 0.5 mW/twice daily; Red light: 1.0 mW/once daily; Red light: 1.0 mW/twice daily; Red light: 2.0 mW/once daily; Red light: 2.0 mW/twice daily
Device: Red LED — In addition to SVS with power for correcting distance refraction, red LED will be performed twice per school day with an interval of at least 4 hours, each treatment last 3 minutes.
  Arms: Red LED: twice daily

SUMMARY:
To explore the minimum power and frequency of Repeated Low-level Red-light (RLRL) to control myopia progression in low-myopic children aged 8-10 years, and the rebound effect of low-myopic children after discontinuation of RLRL with different combinations of power and frequency.

DETAILED DESCRIPTION:
Myopia has emerged as a significant public health concern in East Asia. The excessive elongation of the axial length ( AL)of the eye, particularly as myopia progresses to high myopia, is associated with mechanical stretching and thinning of the choroid and sclera. This can lead to vision-threatening complications such as myopic macular degeneration, macular hemorrhage, retinal detachment, cataracts, and glaucoma. Given the serious consequences of high myopia and its associated complications, early and effective prevention and control of myopia become a primary focus in safeguarding visual health and enhancing quality of life.

In recent years, RLRL holds significant potential as an effective strategy for preventing and controlling myopia in children and adolescents. However, recent researches prompt further questions: Is the current power of RLRL exposure optimal? Can the frequency of exposure be refined? What is the relationship among exposure power, frequency and myopia control? To explore these questions and clarify the effects of various combinations of exposure power and frequency on myopia progression following RLRL therapy, our research group plans to conduct a prospective, double-blind, single-center, randomized controlled clinical trial. This study aims to provide more comprehensive evidence to support this innovative intervention on myopia prevention and control.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 8-10 years old
2. Low myopia: cycloplegic spherical equivalent refractions (SERs) range from -0.50 (inclusive) to -3.00 diopters (D) and astigmatism less than -2.5 D in either eye.
3. signed informed consent and was able to participate in the study

Exclusion Criteria:

1. Secondary myopia, such as a history of retinopathy of prematurity or other neonatal diseases; syndromic myopia with a known genetic disorder or connective tissue disease, such as Stickler syndrome or Marfan syndrome
2. Strabismus or other binocular vision abnormalities
3. Cloudy refractive media: cloudy cornea, cataract or intraocular lens surgery
4. Eye diseases that affect retinal function: macular degeneration, diabetic retinopathy, retinal detachment, glaucoma or ocular hypertension, endophthalmitis, uveitis, optic neuropathy, etc.
5. History of refractive surgery, internal eye surgery, laser therapy, vitreous injection, etc.
6. diabetes, hypertension and other systemic disorders
7. History of use of retinal toxic drugs, such as hydroxychloroquine, etc.
8. Use of orthokeratology, atropine, multifocal frame glasses and other myopia control methods; children who are currently receiving atropine, orthokeratology, multifocal frame glasses and other myopia control treatment, can be enrolled after 2 weeks of treatment.
9. Other reasons considered unsuitable for inclusion by the study physician, including but not limited to other ocular and systemic disease abnormalities

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-04-09 (Estimated); Study Completion 2025-06-09 (Estimated)

PRIMARY OUTCOMES:
The incidence (%) of axial length increase ≤0.05mm after red light for 3 months measured by the IOL master | 1 week, 1, 2, 3 months
  Incidence rate of axial length shortening > 0.05 mm is characterized as the ratio of number of participants with axial length shortening greater than 0.05 mm to the total number.

SECONDARY OUTCOMES:
The incidence rates (%) of cycloplegic spherical equivalent refraction progressing ≥0.00 D after red light for 3 months measured by the autorefractor | 1 week, 1, 2, 3 months
  Refraction with full cycloplegia is performed with an autorefractor. The data on spherical and cylindrical power and axis is automatically extracted from the autorefractor. The spherical equivalent power (D) is calculated as the spherical power (D) plus half of the cylindrical power (D).
Changes of axial length (mm) after discontinuation of red light for 1 months measured by the IOL master | 4 months
  Change of axial length is characterized as the difference between each follow-up visit and baseline values.
Changes of cycloplegic spherical equivalent refraction (D) after discontinuation of red light for 1 months measured by the autorefractor | 4 months
  Change of cycloplegic spherical equivalent refraction is characterized as the difference between each follow-up visit and baseline values.
Incidence (%) of self-reported adverse events by the quesionnaire including but not limited to glare, flash blindness, and afterimages | 1 week, 1, 2, 3, 4 months
  Incidence of self-reported adverse events is the rate of self-reported adverse events over a specified period for all the subjects.
Change in visual acuity (logMAR) measured by the Early Treatment Diabetic Retinopathy Study (ETDRS) logMAR chart | 1 week, 1, 2, 3, 4 months
  Visual acuity change is characterized as the difference between each follow-up visit and baseline values. An ETDRS chart with standard illumination at a distance of 4 meters is used to measure visual acuity.
Changes in choroidal thickness (μm) measured by the swept-source optical coherence tomography and optical coherence tomography angiography | 1 week, 1, 2, 3, 4 months
  Changes in choroidal thickness (μm) are characterized as the difference between each follow-up visit and corresponding baseline values. Indicators include choroidal vascular index, choroidal thickness and so on.
Changes in the amplitudes of waves (mV) measured by the full-filed electroretinogram | 1 week, 1, 2, 3, 4 months
  Changes in the amplitudes of the waves are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by electroretinogram.
Changes in the the latency of waves (ms) measured by the full-filed electroretinogram | 1 week, 1, 2, 3, 4 months
  Changes in the latecy of the waves are characterized as the difference between each follow-up visit and corresponding baseline values which are measured by electroretinogram.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Eye Disease Prevention & Treatment Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared as open data after proper anonymization.